CLINICAL TRIAL: NCT07287605
Title: Evaluating the Impact of Virtual Reality on Mood in Patients Undergoing Magnetic Resonance-Guided Focused Ultrasound for Medication-Refractory Essential Tremor
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 6390
Record Dates: First submitted 2025-11-18; First posted 2025-12-17 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-11

CONDITIONS: Preoperative Anxiety
Keywords: medication-refractory essential tremor; focused ultrasound; virtual reality intervention; MRgFUS; preoperative anxiety

STUDY DESIGN:
Intervention Model Description: Assigning participants to an intervention with VR exposure in order to assess the health outcomes of anxiety levels. Participants are blinded to which of the two possible VR videos they will see.
Who Masked: Participant
Masking Description: Participants are blinded to which of the two possible VR videos they will see.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exposure to Video number 1 (Experimental): Each participant will be randomized to watch Video number 1, 6-minute VR video associated with the study. Participants will be blinded to the type of video. The study will evaluate the impact of the sights and sounds in the video on anxiety levels.
  Interventions: Device: VR headset: video number 1
- Exposure to Video number 2 (Experimental): Each participant will be randomized to watch Video number 2, 6-minute VR video associated with the study. Participants will be blinded to the type of video. The study will evaluate the impact of the sights and sounds in the video on anxiety levels.
  Interventions: Device: VR headset: video number 2

INTERVENTIONS:
Device: VR headset: video number 1 — A 6-minute virtual reality (VR) video that contains sights and sounds that might affect mood. The video is viewed on a Meta Quest 2 (128GB) VR headset with Touch Controllers. Standard preoperative care is provided to all participants.
  Arms: Exposure to Video number 1
Device: VR headset: video number 2 — A 6-minute virtual reality (VR) video that contains sights and sounds that might affect mood. The video is viewed on a Meta Quest 2 (128GB) VR headset with Touch Controllers. Standard preoperative care is provided to all participants.
  Arms: Exposure to Video number 2

SUMMARY:
The primary objective of this randomized study is to evaluate the effect of a virtual reality (VR) video on pre-treatment anxiety levels in individuals undergoing magnetic resonance-guided focused ultrasound (MRgFUS) treatment for medication-refractory essential tremor (ET). Participants will be randomized to view one of two VR videos, and pre-treatment anxiety levels will be compared between groups.

As a secondary objective, the study will compare patient concerns (including claustrophobia, mental preparedness, and fear of pain, as well as any additional concerns identified during the study) between the two randomized groups.

DETAILED DESCRIPTION:
This study will evaluate the effectiveness of a virtual reality (VR) intervention in reducing preoperative anxiety among adults scheduled to undergo magnetic resonance-guided focused ultrasound (MRgFUS) for essential tremor. Sixty adult participants scheduled for MRgFUS will be randomized to view one of two 6-minute immersive VR procedural videos using a headset prior to treatment.

Preoperative anxiety will be assessed using validated self-report instruments, including the Visual Analogue Scale for Anxiety (VAS), the Amsterdam Preoperative Anxiety and Information Scale (APAIS), and the State-Trait Anxiety Inventory - State version (STAI-S). The primary objective is to compare preoperative anxiety levels between the two VR video groups. A secondary objective is to compare patient concerns between groups, including but not limited to claustrophobia, mental preparedness, and fear of pain, as well as any additional concerns identified through patient reporting.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be over the age of 18 and have been approved and consented for MRgFUS thalamotomy for medication-refractory essential tremor
* Subjects must be and willing to give consent and able to attend all study visits and MRgFUS procedure, understanding the associated risks and benefits.
* Participants must be willing or able to complete questionnaires or have someone who can complete them on their behalf.

Exclusion Criteria:

* Patients prone to epileptic seizures and/or sensory issues will be excluded from the study.
* Patients who have previously undergone an MRgFUS procedure (ipsilateral or contralateral to the hemisphere currently being treated) will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-06-19 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Evaluation of Anxiety Levels by Visual Analogue Scale for Anxiety (VAS-A) | Questionnaires will be collected at two time points: 1.Baseline assessment day (two weeks before the MRgFUS procedure), before and after watching the VR video. 2.Treatment day, prior to the MRgFUS procedure.
  Participants will complete questionnaires to establish baseline anxiety levels. A 10-point numeric rating scale displayed horizontally, ranging from 0 = "Not at all anxious" to 10 = "Extremely anxious." Participants mark the number that best represents their current level of anxiety. Higher scores indicate greater anxiety.
Evaluation of Anxiety Levels by Amsterdam Preoperative Anxiety and Information Scale (APAIS) | Questionnaires will be collected at two time points: 1.Baseline assessment day (two weeks before the MRgFUS procedure), before and after watching the VR video. 2.Treatment day, prior to the MRgFUS procedure.
  Participants will complete questionnaires to establish baseline anxiety levels. The Amsterdam Preoperative Anxiety and Information Scale (APAIS) is a 12-item self-administered questionnaire used to assess preoperative anxiety. Each item is rated on a 5-point scale (1 = not at all to 5 = extremely).
  Higher scores indicate greater anxiety or information need. In this study, patient concerns may include anesthesia, head shaving, potential side effects and desire for additional procedural information.
Evaluation of Anxiety Levels by State-Trait Anxiety Inventory - State Subscale (STAI-S) | Questionnaires will be collected at two time points: 1.Baseline assessment day (two weeks before the MRgFUS procedure), before and after watching the VR video. 2.Treatment day, prior to the MRgFUS procedure.
  Participants will complete questionnaires to establish baseline anxiety levels. The State-Trait Anxiety Inventory - State Subscale (STAI-S) is a validated self-report questionnaire used to measure situational ("state") anxiety - how the participant feels "right now, at this moment." Each item is rated on a 4-point scale ranging from 1 = not at all to 4 = very much so. Higher scores indicating greater anxiety.

SECONDARY OUTCOMES:
Participant feedback on the VR experience | Feedback will be collected at two time points: 1.Baseline assessment day (two weeks before the MRgFUS procedure), before and after watching the VR video. 2.Treatment day, prior to the MRgFUS procedure.
  Participants will be asked to provide feedback on the VR experience.
Adverse Effects Associated With Watching the VR Video | Adverse effects will be monitored at two time points: 1.Baseline assessment day (two weeks before the MRgFUS procedure). 2.Treatment day, prior to the MRgFUS procedure.
  Participants will be monitored for any adverse effects experienced during or immediately after viewing the VR video. Reported effects may include, but are not limited to, dizziness, nausea, eye strain, headache, motion sickness, or discomfort related to wearing the VR headset. All adverse effects will be self-reported by participants. The frequency, type, and severity of adverse effects will be recorded and compared between the two randomized VR video groups.

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Jennifer Rabin, PhD, C.Psych, Principal Investigator — Sunnybrook
Locations (1):
- Sunnybrook Health Sciences, North York, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No